CLINICAL TRIAL: NCT04872985
Title: Efficacy and Safety of Pyrotinib in Combination With Neoadjuvant Chemotherapy in Stage II-III HR+/HER2-, HER4 High Expression Breast Cancer Patients: A Phase II, Single-center, Randomized, Double-Blinded, Placebo-Controlled Trial
Brief Title: Pyrotinib Plus Neoadjuvant Chemotherapy in HR+/HER2-, HER4-High Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Erwei Song, M.D., Ph.D., MD.Ph.D., Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MA-BC-II-018
Record Dates: First submitted 2021-04-29; First posted 2021-05-05 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Hormone-receptor Positive Breast Cancer
Keywords: Pyrotinib; Pan-HER TKI; HER4
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; Epirubicin; Cyclophosphamide; Docetaxel; Taxes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Pyrotinib+ AC/EC followed by T (Experimental): 400 mg Pyrotinib orally once per day with four cycles of epirubicin (100 mg/m2) (or doxorubicin hydrochloride liposome injection 30mg/m2) and cyclophosphamide (600 mg/m2) intravenously, once every 3 weeks, followed by four cycles of docetaxel (100 mg/m2) intravenously, once every 3 weeks (or 260mg/m2 nab-paclitaxel once every 3 weeks for 4 cycles, or 12 cycles of weekly nab-paclitaxel 120mg/m2 intravenously). Pyrotinib starts with a dose of 240 mg once daily for one week, followed by 320 mg once daily for the next week, before transitioning to 400 mg once daily as maintenance therapy.
  Interventions: Drug: Pyrotinib; Drug: Epirubicin; Drug: Doxorubicin Hydrochloride Liposome Injection; Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Nab paclitaxel
- Arm 2: Placebo+ AC/EC followed by T (Placebo Comparator): 400 mg placebo orally once per day with four cycles of epirubicin (100 mg/m2) (or doxorubicin hydrochloride liposome injection 30mg/m2) and cyclophosphamide (600 mg/m2) intravenously, once every 3 weeks, followed by four cycles of docetaxel (100 mg/m2) intravenously, once every 3 weeks (or 260mg/m2 nab-paclitaxel once every 3 weeks for 4 cycles, or 12 cycles of weekly nab-paclitaxel 120mg/m2 intravenously) .
  Interventions: Drug: Epirubicin; Drug: Doxorubicin Hydrochloride Liposome Injection; Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Nab paclitaxel; Drug: Placebo

INTERVENTIONS:
Drug: Pyrotinib — 400 mg orally once per day. Pyrotinib starts with a dose of 240 mg once daily for one week, followed by 320 mg once daily for the next week, before transitioning to 400 mg once daily as maintenance therapy.
  Arms: Arm 1: Pyrotinib+ AC/EC followed by T
Drug: Epirubicin — 100 mg/m2,q3W*4
  Other Names: E
Drug: Doxorubicin Hydrochloride Liposome Injection — 30mg/m2, q3w*4
  Other Names: A
Drug: Cyclophosphamide — 600 mg/m2, q3w*4
  Other Names: C
Drug: Docetaxel — 100 mg/m2, q3w*4
  Other Names: T
Drug: Nab paclitaxel — 120mg/m2 qw*12 or 260mg/m2 q3w*4
Drug: Placebo — 400 mg orally once per day
  Arms: Arm 2: Placebo+ AC/EC followed by T

SUMMARY:
This is a Phase II, single-center, double-blind, placebo-controlled, randomized study of Pyrotinib in combination with Doxorubicin/Epirubicin and Cyclophosphamide followed by Docetaxel/nab-Paclitaxel as neoadjuvant therapy for women with hormone receptor positive HER2-negative stage II to III breast cancer. Patients randomized to the study arm/control arm will receive standard neoadjuvant chemotherapy in combination with pyrotinib/placebo, respectively. The primary endpoint of the study is the residual cancer burden 0/I (RCB 0/I) and total pathological complete response (tpCR) rate. Secondary endpoints include the breast pCR (bpCR) rate, objective response rate(ORR), event-free survival (EFS), overall survival (OS), rate of change in the Ki-67 proliferation index, correlations between potential biomarkers and treatment efficacy, and toxicity.

DETAILED DESCRIPTION:
Pyrotinib is an oral, irreversible pan-ErbB receptor tyrosine kinase inhibitor (TKI) with activity against epidermal growth factor receptor HER1(EGFR), HER2 and HER4. Improvement of the chemotherapy efficacy and good tolerability have been shown by several stage II and III clinical trials in both the neoadjuvant and metastasis setting in HER2-positive breast cancers. Yet, the anti-tumor effect of Pyrotinib by targeting HER4 has not been determined. Preclinical studies show that HER4 is relatively highly expressed in hormone receptor positive and HER2-negative(HR+/HER2-) breast cancers. In MCF7 cell lines, Pyrotinib effectively repressed phosphorylation of MAPK and Akt signal transduction pathways to inhibit tumor cell proliferation. In HR+/HER2- tumor xenografts, Pyrotinib has been observed to inhibit tumor growth in a dose-dependent manner (unpublished data). Taken together, the data support the rationale that Pyrotinib may be efficacious in HER4 high expressed HR+/HER2- breast cancer and in combination with chemotherapy may lead to a better RCB 0/I and pCR rate in the neoadjuvant setting.

The study is a two-arm design with a 1:1 allocation ratio (equal numbers of patients randomized to Arms 1, 2). The sample size will be up to 140 patients with about 70 evaluable patients in each arm. Accrual is expected to occur over 48 months. Patients will be randomized to one of the two neoadjuvant therapy regimens: Patients in Arm 1 will be assigned to receive 400 mg Pyrotinib orally once per day with four cycles of epirubicin (100 mg/m2) (or doxorubicin hydrochloride liposome injection 30mg/m2) and cyclophosphamide (600 mg/m2) intravenously, once every 3 weeks, followed by four cycles of docetaxel (100 mg/m2) intravenously, once every 3 weeks(or nab-paclitaxel 260mg/m2 q3w, or 12 cycles of weekly nab-paclitaxel 120 mg/m2) . Dosage reduction of pyrotinib is permitted from 400 mg to 320 mg or 240 mg if Pyrotinib-related AEs are experienced. In Arm 2 (control), Pyrotinib will be replaced by 400mg placebo provided by the same pharmacy company.

In all arms, clinical response will be evaluated by breast MRI. The primary endpoint will be assessed with the paraffin embedded pathological specimens collected from surgery. Submission of tumor samples for the correlative science studies will be optional for all patients. For patients who agree, pathological sections of core biopsy specimen before treatment (after the patient has signed the consent form and has been screened for eligibility) and pathological sections of surgery residual disease specimen after the completion of the treatment are collected. In addition, a blood sample collected after randomization (before the start of study therapy and after the completion of the neoadjuvant therapy) will also be required for the correlative studies.

ELIGIBILITY:
Inclusion Criteria:

* Presenting with histological(by core needle biopsy or by limited incisional biopsy) proven hormone receptor positive (ER≥10% and/or PR ≥1%), HER2 negative(IHC ≤2+ and/or FISH-) , stage II/ III breast cancer.
* Have clinical indication for neoadjuvant therapy.
* HER4 IHC score ≥ 4.
* Measurable disease (breast and/or lymph nodes).
* The Eastern Cooperative Oncology Group (ECOG) performance status must be 0 or 1.
* Adequate bone marrow function (within 4 weeks prior to registration): WBC≥3.0x109/l, neutrophils ≥1.5 x 109/l, platelets ≥100 x 109/l.
* Adequate liver function (within 4 weeks prior to registration): bilirubin ≤1.5 x upper limit of normal (UNL) range, ALAT and/or ASAT ≤2.5 x UNL, Alkaline Phosphatase ≤5 x UNL.
* Adequate renal function (within 4 weeks prior to registration): the calculated creatinine clearance should be ≥50 ml/min.
* Patients must have the ability to swallow oral medication.
* Without history of any kind of treatment to known malignancy (solid tumor or hematologic).
* Written informed consent.
* Accessible for treatment and follow-up.

Exclusion Criteria:

* Evidence of stage IV breast cancer.
* Contralateral invasive breast cancer or Inflammatory breast cancer.
* History of non-breast malignancies (except for in situ cervical cancers, basal cell carcinoma of the skin, squamous cell carcinomas of the skin or thyroid papillary carcinoma that had received curative treatment before enrollment) within 5 years prior to randomization.
* Known metastatic disease from any malignancy (solid tumor or hematologic).
* Serious other diseases as infections (hepatitis B, C and HIV), recent myocardial infarction, clinical signs of cardiac failure or clinically significant arrhythmias or on screening, any of the following cardiac parameters: bradycardia (heart rate <50 at rest) or QTcF ≥450 msec.
* Known hypersensitivity reaction to any of the components of the treatment.
* Pregnancy or lactation at the time of randomization.
* Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or sign meaningful informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
RCB 0/I (Residual cancer burden 0/I) rate | At the time of surgery
  defined as the proportion of patients whose surgical specimens after neoadjuvant therapy were pathologically assessed as RCB 0 or RCB I.
tpCR (total pCR) rate | At the time of surgery.
  ypT0/isN0, number of participants with by no histologic evidence of invasive tumor cells in the surgical breast and axillary specimen.

SECONDARY OUTCOMES:
bpCR (breast pCR) | At the time of surgery.
  ypT0/is, number of participants with by no histologic evidence of invasive tumor cells in the surgical breast specimen.
ORR (objective response) rate | At the time of surgery.
  the percentage of patients with a final overall response of CR or PR relative to the appropriate analysis set. Clinical response will be evaluated by breast MRI.
EFS (event-free survival) at 3 and 5 years | EFS will be determined at 3 and 5 years after randomization
  EFS is defined as the time from randomization to the date of progression(according to RECIST 1.1 ) of disease that precludes surgery, local relapse, regional relapse, distant relapse, second primary invasive breast cancer including contralateral breast cancer, or death due to any cause which ever occurred first.
OS (overall survival) at 3 and 5 years | OS will be determined at 3 and 5 years after randomization
  OS is defined as the time from randomization to date of death.
Rate of change in the Ki-67 proliferation index | Baseline and at the time of surgery
  defined as change of Ki-67 expression in the tumor tissue before and after neoadjuvant therapy
The correlation of potential biomarkers with the RCB 0/I, tpCR, bpCR and ORR rate. | The correlation with RCB 0/I, tpCR, bpCR and ORR will be assessed when the surgery is performed on the last enrolled patients.
  We will used immunohistochemistry (IHC) method to assess the positive percentage of ER, PR, Ki67%, as well as the HER4 scores, and the status EGFR, HER3, and PD-L1 of the specimen from primary core biopsy at baseline. The IHC4 score will be calculated using our modified method (Jin et al. Oncologist. 2020 Aug;25(8):e1170-e1180.). The correlation between these biomarkers with treatment efficacy (RCB 0/I, tpCR, bpCR and ORR) will be explored.
The correlation of potential biomarkers with EFS and OS. | The correlation with EFS and OS will be performed at 5 years after the enrollment of the last patient.
  We will used immunohistochemistry (IHC) method to assess the positive percentage of ER, PR, Ki67%, as well as the HER4 scores, and the status EGFR, HER3, and PD-L1 of the specimen from primary core biopsy at baseline, as well as the residual surgical specimen after neoadjuvant chemotherapy. The IHC4 score will be calculated using our modified method (Jin et al. Oncologist. 2020 Aug;25(8):e1170-e1180.). The correlation between these biomarkers with EFS and OS will be analyzed
AE (Adverse Event) and SAE (Serious Adverse Event) rate | Toxicity will be assessed from start treatment up to 30 days following the last dose of treatment.
  Toxicities are graded according to NCI CTCAE v4.03.
The correlation between NGS sequencing and ctDNA data with clinical outcomes(Optional). | The correlation with pCR will be assessed when the surgery is performed on the last enrolled patients. The correlation with EFS and OS will be performed at 5 years after the enrollment of the last patient.
  NGS sequencing will be performed with the pathological section of primary core biopsy and surgery residual specimen, and the ctDNA will be extracted from the patients' serum at baseline and the date of surgery, if with the agreement of participants. The correlation between these biomarkers with clinical outcomes (pCR and EFS) will be assessed when possible.

CONTACTS AND LOCATIONS:
Overall Officials: Erwei Song, MD.,Phd., Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun-Yat-Sen Memorial Hospital of Sun-Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided